CLINICAL TRIAL: NCT07332988
Title: Effect of Low-Level Light Therapy on Ocular Surface Parameters in Patients With Graves Disease
Acronym: LLLT-Graves
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Timofte Zorila Mihaela Madalina, Principal Investigator, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 598/20.05.2025
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye Disease (DED); Graves Ophthalmopathy
Keywords: DED associated with Graves Ophtalmopaty; DED; Graves; Ophtalmopaty; LLLT; Photobiomodulation
MeSH Terms: conditions — Dry Eye Syndromes; Graves Ophthalmopathy | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, single-masked, parallel-group trial. Eligible participants diagnosed with Graves' disease are randomly assigned in a 2:1 ratio to receive either low-level light therapy (LLLT) or a sham treatment. Interventions are scheduled once per week over a 4-week period. Clinical outcomes are assessed at baseline, after each treatment session, and at 4, 8, 12 and 16 weeks. Participants remain in their assigned group for the duration of the study, with no crossover between groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLLT Group (Experimental): A total of 20 patients will be enrolled and treated as per the classical protocol for dry eye treatment (4 sessions at weekly intervals and 3 monthly follow ups).The treatment was delivered through a wearable mask emitting polychromatic red and near-infrared light, targeting the eyelids and meibomian glands.
  Ocular surface assessments were performed at baseline (before the first treatment), once a week (before each treatment) for 4 weeks, and later on at one month, 2 months and 3 months follow ups to evaluate the effects of LLLT on tear film quality, inflammation, and meibomian gland function.
  Interventions: Device: Low Light Level therapy
- Sham Group (Sham Comparator): A total of 10 patients will be enrolled and treated as per the classical protocol for dry eye treatment (4 sessions at weekly intervals and 3 monthly follow ups). The procedure mimicked the experience of the active LLLT intervention, using the same mask device without activation of the therapeutic light emission. The ocular surface assessments were conducted at the same time points as the active treatment group-baseline, every week for the first month, at 1 month, 2 months and 3 months follow ups to evaluate tear film function, ocular surface condition, and meibomian gland performance.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Sham (No Treatment) — The sham group had undergone a similar procedure using the Eye-light® device (Espansione Group, Italy), as the one described above but in this case the device emits only 30% of the treatment power. Patients had a similar visual and sensory experience of the treatment but without actual biologic effects.
  Each treatment session lasted a total of 15 minutes. It is non-pharmacological, non-contact, and well-tolerated. The light is delivered through closed eyelids, ensuring safety and comfort. This approach allowed for masking of participants and investigators to minimise bias, while ensuring that patients in the control group received no active therapeutic exposure.
  Arms: Sham Group
Device: Low Light Level therapy — The intervention consists of non-invasive periocular photobiomodulation using the Eye-light® device (Espansione Group, Italy), which delivers low-level polychromatic red and near-infrared light through a specially designed mask. The LLLT mask consisted of light emitting diodes (LEDs) with red light, 633 nm wavelengths. The treatment is designed to improve tear film stability, stimulate meibomian gland activity, reduce ocular surface inflammation. This protocol targets cellular mitochondrial activity to enhance tissue repair and anti-inflammatory effects. Each treatment session lasted a total of 15 minutes. It is non-pharmacological, non-contact, and well-tolerated. The light is delivered through closed eyelids, ensuring safety and comfort, and the device used is CE-marked for ophthalmic applications.
  Arms: LLLT Group

SUMMARY:
This prospective, interventional, randomized, controlled, double-blind clinical study evaluates the effect of Low-Level Light Therapy (LLLT) delivered by a polychromatic periocular mask (Eye-light®️) versus a sham device in adults with dry eye disease (DED) associated with Graves' ophthalmopathy, refractory to conventional topical treatment. The LLLT protocol applies photobiomodulation to eyelid and periocular tissues to support meibomian gland function and reduce tear inflammatory biomarkers. The primary endpoint is the change in tear film stability measured by Non-Invasive Tear Break-Up Time (NIBUT) and Fluorescein Tear Break-Up Time (FBUT). Secondary outcomes include symptom scores (OSDI), Schirmer I test, tear osmolarity, ocular surface staining scales, automated conjunctival hyperemia, blink analysis, meibomian gland morphology (meibography/meiboscale), tear inflammatory biomarkers, and safety/tolerability.

DETAILED DESCRIPTION:
This randomized, single-masked, parallel-group clinical trial was conducted to evaluate the efficacy and safety of low-level light therapy (LLLT) in the management of dry eye disease (DED) in patients diagnosed with Graves Ophthalmopathy. The study was carried out at the Department of Ophthalmology of Clinical Hospital CF Iaşi, Romania, University of Medicine and Pharmacy "Grigore T. Popa" (Iași, Romania), in accordance with the Declaration of Helsinki and ICH-GCP guidelines.

Dry eye disease is a multifactorial disorder characterized by tear film instability and ocular surface inflammation. Patients with Graves' ophthalmopathy often experience a severe form of dry eye that is resistant to conventional topical treatments, resulting in a need of finding new therapies to stabilize the tear-film.

LLLT is a non-invasive photobiomodulation technique that delivers low-intensity, polychromatic red and near-infrared light to target mitochondrial cytochromes and promote cellular activity. Its application in ophthalmology has shown potential to improve meibomian gland function, enhance tear film stability, and downregulate inflammatory cytokines on the ocular surface. However, its utility in patient with diagnosed DED associated with Graves Ophthalmopathy has not been formally evaluated.

Eligible participants included consecutive adults (≥18 years) diagnosed with DED associated with Graves Ophthalmopathy that are refractory to conventional dry eye treatments. Key exclusion criteria were pregnant or breastfeeding patients, uncontrolled systemic disease (other than Graves Disease), use of general corticosteroids in the last 6 months, ocular and orbital surgery in the last 6 months, use of contact lenses in the last month and any active ocular infection or allergy.

Eligible participants were randomly assigned to each the active low-level light treatment group or the sham-control group with the Eye-light unit (Espansione Group Ltd, Funo, Italy). Randomization was performed using a computerized allocation sequence (http://www.sealedenvelope.com). Allocation concealment was ensured through sequentially numbered, opaque, sealed envelopes. Both participants and investigators responsible for clinical evaluations remained unaware of group assignment throughout the study period.

Participants were randomized into two groups: the intervention group received LLLT using the Eye-light® device (Espansione Group, Italy), and the control group received sham treatment with an identical, inactive device. Each treatment session lasted a total of 15 minutes. The LLLT masks consisted of light emitting diodes (LEDs) with red light, 633 nm wavelengths. Participants attended a total of seven visits. The first 4 visits comprised of treatment sessions, each session separated by 1 week. The next 3 visits comprised of a follow-up assessment, 1 month following the final treatment session, 60±7 days after the last treatment and 90±7 days after the last treatment, targeting the periocular region and meibomian glands.

Clinical assessments were performed at baseline (T0), before first mask session, 7 days after T0 (T1), 7 days after T1 (T2), 7 days after T2 (T3), 30±4 days after T3 (T4), 60±7 days after T4 (T5) and 90±7 days after T5 (T6), and included:

1. Tear Collection Procedure: Tear samples were collected using Schirmer type I strips without topical anesthesia to assess changes in tear inflammatory biomarkers using Luminex Human Discovery Assay 9 plex- CD 27, CD 40, ICAM 1, IL 1 beta, IL 10 , MMP8, TNF alfa, TNF RI, TRAIL R2 in patients with Graves' ophthalmopathy . The strips were placed in the lower conjunctival fornix for up to 5 minutes, then individually stored in sterile microtubes at -80 °C.
2. Tear Protein Extraction: For protein extraction, the strips were thawed and incubated in 400 μL of 1.5 M Tris-HCl buffer (pH 8.8) containing protease inhibitors for 3 hours, followed by centrifugation at 16,000× g for 15 minutes (4 °C). Total protein content was determined by Nanodrop (ThermoFischer Scientific), and tear cytokines and chemokines were quantified using a multiplex bead-based immunoassay (R&D Systems) on a Luminex FlexMap3D platform.
3. Analysis Method: Tear proteins will be analyzed using the Luminex® multiplex immunoassay, as recommended by the manufacturer.
4. Clinical Measurements: Ocular Surface Disease Index (OSDI) scores, Schirmer 1 test, number of total blinks in 30s and number of partial blinks within that timeframe, tear meniscus height, subjective lipid layer pattern grading, automated bulbar conjunctival and limbal hyperemia (DEA 520), fluorescein corneal staining and fluorescein staining using the Oxford scale, tear osmolarity and meibography drop-out graded with the meiboscale for upper and lower eyelids, will be measured at each session (T0-T6).

The primary outcome was the change in tear film stability (NIBUT and FBUT) from baseline to 3 months post treatment. Secondary outcomes included all objective ocular surface parameters. Safety was evaluated by monitoring treatment-emergent adverse events and assessing patient tolerability of the device.

Statistical analysis was performed using SPSS (version 30.0.0.0, SPSS Inc., Chicago, IL, USA). The normality of data was evaluated using the Shapiro-Wilk test. For normally distributed variables, repeated measures ANOVA followed by Dunnett's post-hoc tests were used. For non-normally distributed data, the Friedman test with Dunn's correction was applied. A p-value < 0.05 was considered statistically significant.

This is the first prospective study to investigate LLLT in the diagnosed DED associated with Graves Ophthalmopathy patients. The findings aim to provide evidence for integrating non-pharmacological interventions in ocular surface optimization for this category of patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with dry eye disease, particularly associated with Graves' ophthalmopathy.
* Refractory to conventional dry eye treatments (e.g., artificial tears, cyclosporine, corticosteroid eye drops).
* Adult patients (over 18 years old).

Exclusion Criteria:

* Pregnant or breastfeeding.
* Uncontrolled systemic diseases (other than Graves' disease).
* Use of general corticosteroids in the last 6 months.
* Ocular or orbital surgery in the last 6 months.
* Use of contact lenses within the last week.
* Active ocular infection or allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Changes in tear film stability (NIBUT and FBUT) from baseline during the treatment and in the follow-up period in patients with Graves' ophthalmopathy who undergo low-level light therapy (LLLT) | Before first mask session, and weekly before each treatment to the final treatment, at 1 month, 2 months and 3 months follow ups after the final treatment.
  Noninvasive Tear Break-Up Time (NIBUT) is an eye test measuring the stability of the tear film without using dye (fluorescein), making it more accurate than standard tests. It determines how long the tear film stays intact before breaking, with results typically indicating dry eye if the time is under 10 seconds.
  Fluorescein Breakup Time (FBUT) is a diagnostic test measuring the time (in seconds) between the last blink and the appearance of the first dry spot or break in the tear film. Both of these measurements were assessed objectively on average of three repeats in order to obtain the average value using the DEA 520 Dry Eye Analyzer; Moptim / Shenzhen Certainn Technology Co., Ltd., China.
  The primary outcome is the change in the tear film stability from baseline to 3 months after the final treatment, comparing the LLLT group to the sham group.

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | Before first mask session, and weekly before each treatment to the final treatment, at 1 month, 2 months and 3 months follow ups after the final treatment.
  The Ocular Surface Disease Index (OSDI) is a validated 12-item questionnaire used to assess the severity of dry eye symptoms and their impact on vision-related functioning. The total score ranges from 0 to 100, with higher scores indicating greater symptom severity. Participants will complete the OSDI questionnaire at baseline and after every treatment including follow ups. The secondary outcome is the change in total OSDI score from baseline to 3 months after the final treatment, comparing the LLLT group to the sham group.
Schirmer I Test | Before first mask session, and weekly before each treatment to the final treatment, at 1 month, 2 months and 3 months follow ups after the final treatment.
  The Schirmer I Test is a standard diagnostic tool used to measure aqueous tear production. Without anesthesia, a sterile paper strip is placed in the lower conjunctival sac for 5 minutes, and the length of the moistened area (in millimeters) indicates tear secretion. Lower values reflect aqueous-deficient dry eye. The secondary outcome is the change in tear production from baseline to 3 months after the final treatment, comparing results between patients treated with low-level light therapy (LLLT) and those receiving sham treatment.
Tear osmolarity | Before first mask session, at 1 month and 3 months follow ups after the final treatment.
  Tear osmolarity is the measurement of the concentration of solutes (primarily salts) in the tear film, typically expressed in mOsm/L. It serves as a key biomarker for diagnosing and managing dry eye disease (DED), as levels above 308-310 mOsm/L indicate hyperosmolarity (high salt concentration) due to water evaporation or reduced tear production. The secondary outcome is the change in tear osmolarity values from baseline to 3 months after the final treatment, comparing the LLLT group to the sham group.
Tear meniscus height | Before first mask session, and weekly before each treatment to the final treatment, at 1 month, 2 months and 3 months follow ups after the final treatment.
  The tear meniscus height (TMH) is defined as the vertical distance of the collection of tears that accumulates along the margin of the lower eyelid. This measurement is a key clinical index used to non-invasively assess the tear film volume in the eye, primarily for the diagnosis and management of dry eye disease (DED). The secondary outcome is the change in tear meniscus height score from baseline to 3 months after the final treatment, comparing the LLLT group to the sham group.
Meibography graded with the meiboscale for upper and lower eyelids | Before first mask session, and weekly before each treatment to the final treatment, at 1 month, 2 months and 3 months follow ups after the final treatment.
  Meibography is a non-invasive imaging technique that uses infrared light to visualize, capture, and analyze the structure and morphology of the meibomian glands within the eyelids. It is used to diagnose Meibomian Gland Dysfunction (MGD) by identifying gland atrophy, blockages, or loss, which contributes to dry eye syndrome. The secondary outcome is the change in aspect of the meibomian glands from baseline to 3 months after the final treatment, comparing the LLLT group to the sham group
Fluorescein corneal staining | Before first mask session, and weekly before each treatment to the final treatment, at 1 month, 2 months and 3 months follow ups after the final treatment.
  Fluorescein corneal staining is a diagnostic eye test using a fluorescent orange dye and cobalt blue light to highlight damaged, scratched, or diseased areas of the cornea. The dye stains epithelial defects, which glow bright green under the light. It is commonly used to detect foreign bodies, abrasions, ulcers, and dry eye severity. The severity is graded using the Oxford scale (0-5), with higher scores indicating extensive corneal damage. The secondary outcome is the changes in corneal staining aspect from baseline to 3 months after the final treatment, comparing the LLLT group to the sham group
Lipid layer pattern grading | Before first mask session, and weekly before each treatment to the final treatment, at 1 month, 2 months and 3 months follow ups after the final treatment.
  Lipid layer pattern grading is used to subjectively assess the thickness and quality of the tear film's outermost lipid layer. The secondary outcome is the change in the lipid layer from baseline to 3 months after the final treatment, comparing the LLLT group to the sham group
Blinking rate | Before first mask session, and weekly before each treatment to the final treatment, at 1 month, 2 months and 3 months follow ups after the final treatment.
  Blinking rate is defined as the frequency of involuntary, spontaneous eye closures, supporting tear film distribution and ocular surface lubrication, cleansing ad protection. In this study, blinks are recorded over 30s and reported as both complete and incomplete (partial) blinks. The secondary objective is to assess the difference between the quality of blinking (complete/incomplete blinks) from baseline to 3 months after the final treatment, comparing the LLLT group to the sham group.
Automated hyperemia assessment | Before first mask session, and weekly before each treatment to the final treatment, at 1 month, 2 months and 3 months follow ups after the final treatment.
  Automated hyperemia assessment is a method that uses computer software and image processing techniques to objectively and quantitatively measure the level of redness in the conjunctiva (the white part of the eye) from digital photographs. This automation aims to replace traditional, subjective clinical grading scales. The secondary outcome is to assess the improvement of hyperemia from baseline to 3 months after the final treatment, comparing the LLLT group to the sham group.
Tear Inflammatory and Reparative Biomarkers | At baseline and 3 months after the last treatment.
  Tear biomarkers were quantified using a customized Luminex multiplex assay enabling the simultaneous measurement of CD 27, CD 40, ICAM 1, IL 1 beta, IL 10 , MMP8, TNF alfa, TNF RI, TRAIL R2 , in accordance with the manufacturer's recommendations. Briefly, thawed tear samples were diluted 1:2 using the supplied sample diluent. Lyophilized analyte standards were reconstituted with calibrator diluent and combined to generate the highest concentration standard, followed by a three-fold serial dilution to obtain 6 standard points. The measurable concentration ranges for the biomarkers included in the Luminex Human Discovery 9-Plex panel are as follows: CD27 (TNFRSF7) 103-25,000 pg/mL, CD40 Ligand (TNFSF5) 206-50,000 pg/mL, ICAM-1 (CD54) 3,200-775,000 pg/mL, IL-1 beta (IL-1F2) 17.7-4,300 pg/mL, IL-10 4.1-100 pg/mL, MMP-8 226-55,000 pg/mL, TNF-alpha 8.23-2,000 pg/mL, TNF RI (TNFRSF1A) 49.4-12,000 pg/mL, and TRAIL R2 (TNFRSF10B) 20.6-5,000 pg/mL. The data acquisition carried out on a Luminex.
Clinical Activity Score (CAS) | At baseline (before treatment), 1 month and 3 months follow up.
  The Clinical Activity Score (CAS) is a 7-point, binary checklist used to measure active inflammation in Thyroid Eye Disease (TED/Graves' orbitopathy). A score of (>3) indicates active, often immunosuppressive-responsive disease. It assesses seven key signs: spontaneous pain, gaze pain, lid swelling, lid redness, conjunctival injection, chemosis, and caruncle inflammation. The secondary outcome is the change in the clinical activity score from baseline to 1 month and 3 months follow ups after the final treatment, comparing the LLLT group to the sham group.
Exophthalmometry | At baseline (before treatment), 1 month and 3 months follow up.
  Exophthalmometry is a non-invasive clinical technique used to quantify the forward protrusion (proptosis) of the eyeball relative to the lateral orbital rim, measured in millimeters. It is used to monitor conditions like thyroid eye disease.
  The secondary outcome is the change in the exophthalmometry from baseline to 1 month and 3 months follow ups after the final treatment, comparing the LLLT group to the sham group.

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Madalina Timofte Zorila, Principal Investigator — University of Medicine "Gr. T. Popa", Iasi, Romania
Locations (1):
- University of Medicine and Pharmacy "Grigore T. Popa", Iași, Iaşi, Romania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including demographics (age, sex), baseline and follow-up ocular surface measures, including BUT, Schirmer I test, tear osmolarity, ocular surface staining scales, automated conjunctival hyperemia, blink analysis, meibomian gland morphology, tear inflammatory biomarkers, and thyroid-related clinical scores and biomarkers. No personally identifiable information will be shared. Data will be provided upon reasonable request for ethics/IRB-approved research purposes only.
Supporting Information: Study Protocol, ICF, CSR